CLINICAL TRIAL: NCT04571177
Title: Developing PET Perfusion Imaging Techniques and Comparing Them to CT Perfusion Imaging in Stroke Patients
Brief Title: PET Perfusion Imaging Techniques and Comparing Them to CT Perfusion Imaging in Stroke
Status: Active, not recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Version 1.0 28AUG2019
Record Dates: First submitted 2020-05-19; First posted 2020-09-30 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adult patients who are diagnosed with an acute supratentorial ischemic stroke within 48 hrs of onset will be enrolled into the study. Participants will undergo both a CT Scan and PET scan within 7 days of onset. Participants will have the option to undergo a second PET scan with fluorodeoxyglucose (FDG).

DETAILED DESCRIPTION:
Patients older than 18 years of age diagnosed with an acute supratentorial ischemic stroke within 48 hrs of symptom onset will be prospectively enrolled. Research imaging will be obtained before 7 days after symptom onset. The patient will receive the standardized treatment protocol at the hospital. Informed consent will be obtained from each patient or a substitute decision maker for each individual imaging study (CTP, Rb PET, and FDG PET). The patient will be given the option of undergoing the CTP imaging with the Rb PET only or both the Rb PET and FDG PET components.

ELIGIBILITY:
Inclusion Criteria:

* Age: >18 yo
* Gender: male or female
* Acute (within 7 days from symptom onset) Supratentorial Ischemic Stroke

Exclusion Criteria:

* 1) Planned surgical intervention
* 2) Severely abnormal blood glucose level (will be excluded from FDG PET imaging)
* 3) Unable to undergo CTP or PET imaging (i.e. claustrophobia)
* 4) Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are older than 18 years of age diagnosed with an acute supratentorial ischemic stroke within 48 hrs of onset will be enrolled into the study. Both male and female patients will be enrolled. We want diversity among participants in order to gain insightful information about acute supratentorial ischemic stroke as possible. A broad range in age, along with enrolling both male and female participants will allow greater diversity.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare PET brain perfusion imaging to CTP | through study completion, 1 year from start of recruitment
  Imaging of CTP images with the Rb PET only or both the Rb PET and FDG PET with CTP imaging components to evaluate blood flow and metabolism mismatches.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Buck, Principal Investigator — Associate Professor
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided